CLINICAL TRIAL: NCT06929130
Title: Refractive and Topographic Changes After Strabismus Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Mohammed Moawad Ahmed, residant doctor, Assiut University
Other Study IDs: Ref&TopgraphStrabismus Surg
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Strabismus Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group: patients diagnosed with concomitant strabismus requiring surgical correction

SUMMARY:
Strabismus, characterized by a misalignment of the eyes, is a common condition that can result in functional and cosmetic issues, often affecting vision and binocular coordination. Strabismus surgery aims to correct the alignment by adjusting the extraocular muscles, but while the primary goal of surgery is to restore ocular alignment, refractive changes may occur as a secondary effect (1).

The traditional view of strabismus surgery is that it is more difficult to plan than to perform. Nevertheless, some complications sometimes have some clinical significance and may affect the visual acuity, physical appearance, and future life of the patients (2).

Refractive changes are among the complications of strabismus surgery. This is mostly attributed to the fact that surgical interventions to the extraocular muscles change the vectorial forces transmitted to the cornea via the scleral pathway (3).

Other theories on this subject include postoperative scleral wound healing, edema in the orbit and eyelids, change in ciliary body blood flow, and change in crystalline lens shape and curvature. In addition, if the anterior ciliary arteries are damaged during strabismus surgery, the supply of the anterior segment may be disrupted and changes in parameters may occur accordingly (4).

Also, surface tension changes in adjacent tissues due to changes in muscle tension after surgery may result in changes in corneal and anterior segment measurements (5).

The timing of refractive changes after surgery also varies. Some patients experience changes in their refractive status shortly after surgery, while others may develop these changes months or even years later. This delayed onset can make it more challenging to identify the precise cause of the refractive shift, as it may not always be immediately apparent following the initial surgical correction (6).

Research shows that post-strabismus surgery can result in myopic shifts, especially in patients with esotropia, and hyperopic shifts in exotropia. Astigmatism can also develop due to corneal shape changes. Preexisting refractive errors, age, strabismus type, surgical technique, and surgeon experience also influence post-surgical changes .

To investigate the refractive changes that occur following strabismus surgery, with a focus on identifying the type and timing of refractive shifts (such as myopia, hyperopia, or astigmatism) and their association with the type of strabismus and surgical technique used.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with concomitant strabismus requiring surgical correction.
* Clear ocular media.

Exclusion Criteria:

* Patients with significant ocular pathology (e.g., cataracts, glaucoma,posterior segment pathology).
* Patients who have undergone previous intraocular or strabismus surgeries.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with concomitant strabismus requiring surgical correction.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
refractive error | 6 month
  spherical equivalent of refractive error (measured in diopters, D) before and after strabismus surgery at different follow-up intervals